CLINICAL TRIAL: NCT05124860
Title: A Longitudinal Investigation of Energy Expenditure and Substrate Utilization in Critically Ill Patients: a Prospective Observational Multi-center Study
Brief Title: A Longitudinal Investigation of Energy Expenditure and Substrate Utilization in Critically Ill Patients
Acronym: EPIC
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Martin Sundstrom Rehal, Principal Investigator, Karolinska University Hospital
Other Study IDs: K 2021-6909
Record Dates: First submitted 2021-10-25; First posted 2021-11-18 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Critical Illness
Keywords: Energy expenditure; Indirect calorimetry; Metabolism; Prolonged critical illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Indirect calorimetry — Measurement of metabolic rate (kcal/day) by respiratory gas analysis.

SUMMARY:
The metabolic alterations associated with critical illness have significant implications for the nutritional management of ICU patients. Despite this, little is known about these changes in patients requiring prolonged organ support and nutritional therapy.

The overall aim of this study is to describe changes in metabolism over time in a large prospective cohort of patients requiring >10 days of ICU care. Our hypothesis is that there is a significant change in mean energy expenditure and respiratory quotient (RQ) between the early (day 1-3), intermediate (day 4-10) and late (>10 days) phase in ICU.

DETAILED DESCRIPTION:
Background

Critical illness has profound effects on human metabolism. The most prominent feature in the early phase is an upregulation of catabolic pathways, which promotes the production of endogenous energy substrates and net protein breakdown [1].

There is very little published data describing trends of energy expenditure and substrate utilization in patients with a prolonged ICU stay. While this group only constitutes a small fraction of ICU patients, it accounts for a large part of ICU resource allocation, morbidity and mortality [2]. Several studies have been conducted in recent years to better characterize patients with persistent critical illness, focusing on markers of catabolism and inflammation [3, 4]. It is not known if these changes are associated with alterations in energy metabolism and substrate utilization.

Bridging these knowledge gaps will improve our understanding of the nutritional needs and metabolism of patients beyond the early phase in ICU. We therefore plan to conduct a prospective observational multi-center study to address these questions.

Aim and hypothesis

The overall aim of this project is to describe longitudinal changes in energy expenditure and associated clinical characteristics in a large cohort of patients with a prolonged ICU stay. Our hypothesis is that there is a significant change in mean energy expenditure and respiratory quotient (RQ) between the early (day 1-3), intermediate (day 4-10) and late (>10 days) phase in ICU. Correlations between metabolic rate and other clinical characteristics will also be analysed for hypothesis-generating purposes.

Population

All adult ICU patients with at least one measurement of energy expenditure by indirect calorimetry at participating study sites will be included in the study. Study sites are encouraged to routinely perform indirect calorimetry every 3-4 days. Study subjects will be followed until ICU discharge or death, whichever comes first.

Data collection and reporting

Patient data will be reported pseudonymized through a secure online form.

On admission

* Admission date
* Admission diagnosis (ICD-10)
* Surgery prior to admission (YES/NO), elective or emergent
* Outcome prediction score (SAPS 3, APACHE III/IV, MPM, etc.) and risk of death on admission (%)
* ICU source admission (ER/ward/OT/other ICU)
* Days in hospital before ICU admission

Demographic and anthropometric data:

* Sex (male/female)
* Age (years)
* Weight (kg)
* Height (cm)

Chronic comorbidities registered in electronic health records (YES/NO):

* Hypertension
* Ischemic heart disease
* Heart failure
* Diabetes mellitus
* COPD
* Chronic kidney disease
* End-stage renal disease
* Liver cirrhosis
* Active cancer (not in complete remission)
* Haematological malignancy
* Solid organ transplant

On the day of each indirect calorimetry

* REE (kcal/24 h), RQ, VO2 (ml/min), VCO2 (ml/min) and date of investigation
* Invasive mechanical ventilation (YES/NO) or renal replacement therapy (YES/NO)

If YES to invasive mechanical ventilation:

* Fraction of inspired oxygen
* Positive end-expiratory pressure (cmH2O)

Factors that may influence REE:

* Sequential organ failure assessment (SOFA) score
* Fever (≥38.5 ℃) within 2h of measurement (YES/NO/MISSING)
* Richmond Agitation-Sedation Scale score

Results of daily blood tests if available from routine testing:

* P-CRP (mg/L)
* P-albumin (g/L)
* P-urea (mmol/L)
* P-creatinine (μmol/L)
* Haemoglobin (g/L)

Medications, nutrition and other therapies:

* Infusions of vasoactive medications (YES/NO, if YES → name of medication(s))
* Infusions of sedatives or analgesics (YES/NO, if YES → name of medication(s), if propofol → infusion rate at time of measurement)
* Infusions of parenteral and/or enteral nutrition (YES/NO, if YES → brand name, formulation and rate at time of measurement)

On discharge

* Discharge date
* Survival status (ALIVE/DEAD)
* Sepsis during ICU stay (NO/SEPSIS/SEPTIC SHOCK)

Sample size considerations

The goal of this study is to include ≥200 patients with an ICU length of stay of >10 days. Based on data from the Swedish Intensive Care Registry between 2015-2019, these patients accounted for 5% of all ICU admissions [5]. This proportion is comparable to results from a registry study conducted in Australia and New Zealand of over one million ICU admissions [2]. Based on these figures we intend to screen 6000 unique patients for study participation, accounting for the possibility that multiple measurements of indirect calorimetry are not consistently performed. In total we expect to include around 1250 unique subjects with at least one measurement with indirect calorimetry.

Statistics

Descriptive data will be presented as mean +/- standard deviation or median (interquartile range) as appropriate. The primary and secondary outcome measures will be analysed using a generalized linear mixed-effects model. Exploratory outcomes and their association to other clinical variables will be analysed using generalized linear regression models. If values are found to be not missing at random, conditional logistic regression censoring will be used to calculate inverse probability weights for accounting for difference in drop-out probabilities.

ELIGIBILITY:
Inclusion Criteria:

1. >/= 18 years old.
2. Admitted to the ICU of a participating study site.
3. At least one measurement of energy expenditure performed during ICU stay.

Exclusion Criteria:

1. Patients readmitted to the ICU of a participating study site >72 hours after ICU discharge and already included in the study (≥1 measurement of energy expenditure performed during prior admission). If a patient is readmitted within ≤72 hours of ICU discharge this is considered a continuation of the last ICU admission for the purposes of this study.
2. Burns >20% of body surface area.
3. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult intensive care unit patients with ≥1 measurement of energy expenditure by indirect calorimetry.
Sampling Method: Non-Probability Sample
Enrollment: 714 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Change in resting energy expenditure over time in patients who stay in ICU for >10 days. | From date of ICU admission to the date of ICU discharge or death, whichever came first, assessed up to 24 months.
  Kcal/kg adjusted body weight/24 hours.

SECONDARY OUTCOMES:
Change in respiratory quotient over time in patients who stay in ICU for >10 days. | From date of ICU admission to the date of ICU discharge or death, whichever came first, assessed up to 24 months.
  Quotient of carbon dioxide production and oxygen consumption.
Change in resting energy expenditure (kcal/kg/day) over time in patients who stay in ICU for ≤10 days. | From date of ICU admission to the date of ICU discharge or death, whichever came first, assessed up to 24 months.
  Kcal/kg adjusted body weight/24 hours.
Change in respiratory quotient over time in patients who stay in ICU for ≤10 days. | From date of ICU admission to the date of ICU discharge or death, whichever came first, assessed up to 24 months.
  Quotient of carbon dioxide production and oxygen consumption.

OTHER OUTCOMES:
Correlations between energy expenditure/respiratory quotient and markers of inflammation, protein catabolism, antecedent characteristics and outcomes. | From date of ICU admission to the date of ICU discharge or death, whichever came first, assessed up to 24 months.
  CRP, albumin, urea/creatinine ratio, age, sex, SOFA, ICU mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sundström Rehal, MD PhD, Principal Investigator — Karolinska University Hospital; Olav Rooyackers, PhD, Study Chair — Karolinska Institutet
Locations (7):
- Australia (2):
  - Royal Melbourne Hospital, Melbourne
  - The Alfred, Melbourne
- Gelderse Vallei Hospital, Ede, Netherlands
- Sweden (3):
  - Karolinska University Hospital, Huddinge, Stockholm County
  - Universitetssjukhuset Örebro, Örebro
  - Capio S:t Görans Sjukhus, Stockholm
- Lucerne Cantonal Hospital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Preiser JC, Ichai C, Orban JC, Groeneveld AB. Metabolic response to the stress of critical illness. Br J Anaesth. 2014 Dec;113(6):945-54. doi: 10.1093/bja/aeu187. Epub 2014 Jun 26. PMID 24970271
- [Background] Iwashyna TJ, Hodgson CL, Pilcher D, Bailey M, van Lint A, Chavan S, Bellomo R. Timing of onset and burden of persistent critical illness in Australia and New Zealand: a retrospective, population-based, observational study. Lancet Respir Med. 2016 Jul;4(7):566-573. doi: 10.1016/S2213-2600(16)30098-4. Epub 2016 May 4. PMID 27155770
- [Background] Haines RW, Zolfaghari P, Wan Y, Pearse RM, Puthucheary Z, Prowle JR. Elevated urea-to-creatinine ratio provides a biochemical signature of muscle catabolism and persistent critical illness after major trauma. Intensive Care Med. 2019 Dec;45(12):1718-1731. doi: 10.1007/s00134-019-05760-5. Epub 2019 Sep 17. PMID 31531715
- [Background] Nakamura K, Ogura K, Nakano H, Naraba H, Takahashi Y, Sonoo T, Hashimoto H, Morimura N. C-reactive protein clustering to clarify persistent inflammation, immunosuppression and catabolism syndrome. Intensive Care Med. 2020 Mar;46(3):437-443. doi: 10.1007/s00134-019-05851-3. Epub 2020 Jan 9. PMID 31919541
- See also: Reporting on length of ICU stay 2015-2019 from the Swedish ICU Registry database. — https://portal.icuregswe.org/utdata/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT05124860/Prot_SAP_002.pdf